CLINICAL TRIAL: NCT00003794
Title: Quality of Life in Ovarian Germ Cell Cancer Survivors
Brief Title: Quality-of-Life Study of Patients With Previously Treated Ovarian Cancer
Status: Terminated | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Other Study IDs: CDR0000066937; GOG-9901
Record Dates: First submitted 1999-11-01; First posted 2003-10-29 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2005-11

CONDITIONS: Ovarian Cancer
Keywords: stage I ovarian germ cell tumor; stage II ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Quality-of-life assessment of patients undergoing cancer treatment may help determine the intermediate- and long-term effects of treatment in patients with cancer.

PURPOSE: This clinical trial studies the quality of life in patients with previously treated ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare quality of life in terms of health status, sexual functioning, psychological/emotional well being, and social functioning in ovarian germ cell cancer survivors vs a matched healthy control group. II. Predict quality of life in these patients through the additive effects of cancer diagnosis and treatment, sociodemographic characteristics, other stressors, and social network variables.

OUTLINE: Patients identify up to 3 healthy acquaintance controls within 3 years of the same age. Patients and controls complete a written questionnaire, which takes about 30 minutes, and a telephone interview, which takes about 1 hour, to assess quality of life.

PROJECTED ACCRUAL: A total of 190 patients and 190 healthy controls will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: History of early or advanced ovarian germ cell tumors Continuously disease free for at least 2 years prior to study Must have been enrolled on GOG protocols 45, 78, 90, and 116 or similar protocols of cisplatin-based chemotherapy at M.D. Anderson Cancer Center

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Must be able to complete a written questionnaire and telephone interview in English

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Primary Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Williams, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (4):
- United States (4):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Monahan PO, Champion VL, Zhao Q, Miller AM, Gershenson D, Williams SD, Cella D. Case-control comparison of quality of life in long-term ovarian germ cell tumor survivors: a gynecologic oncology group study. J Psychosoc Oncol. 2008;26(3):19-42. doi: 10.1080/07347330802115715. PMID 19042263
- [Result] Williams SD, Miller AM, Cella D, et al.: Relationship issues and sexual functioning in ovarian germ cell cancer survivors. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-845, 2001.